CLINICAL TRIAL: NCT05606289
Title: A Randomized, Controlled Trial of Crisis Intervention Team (CIT) Mental Health Training for Police Officers
Brief Title: Trial of Crisis Intervention Team (CIT) Mental Health Training for Police Officers
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University of Wisconsin, Milwaukee (Other); Research Foundation for Mental Hygiene, Inc. (Other); Wayne State University (Other)
Responsible Party: Principal Investigator, Michael Compton, Professor of Psychiatry, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 8378; R01MH128500 (NIH)
Record Dates: First submitted 2022-10-24; First posted 2022-11-04 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Officers' Skills and Behaviors
Keywords: Crisis Intervention Team (CIT); Police Officers; Mental Health
MeSH Terms: conditions — Behavior; Psychological Well-Being | interventions — serum P-component

STUDY DESIGN:
Intervention Model Description: Single-blind, parallel-group RCT
Who Masked: Outcomes Assessor
Masking Description: The investigators will blind the rater, who would code the video-recorded outcome behaviors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CIT officers (Experimental): Police officers randomized to the experimental group will receive a 40-hour CIT training curriculum.
  Interventions: Behavioral: Crisis Intervention Team (CIT) training
- Non-CIT officers (No Intervention): Police officers randomized to the no-intervention group will not receive the 40-hour CIT training curriculum.

INTERVENTIONS:
Behavioral: Crisis Intervention Team (CIT) training — Standard 40-hour CIT training given in one week.
  Other Names: CIT mental health training
  Arms: CIT officers

SUMMARY:
The goal of this clinical trial is to learn the effect, or lack thereof, of the Crisis Intervention Team (CIT) training among police officers. The main questions it aims to answer are:

* Whether the 40-hour CIT training improves police officers' verbal crisis de-escalation skills / non-verbal physical behavior
* Whether police officers with and without CIT training use different procedural justice and make different disposition-related decisions

Participants will:

* Receive or not receive CIT training depending on whether they are randomized to the intervention group or the control group.
* Participate in three assessments: baseline before the randomization, 3-months post-randomization, and 6-month post-randomization.

Researchers will compare police officers who were randomized to the control group with police officers who were randomized to the intervention group to see if receiving the CIT training make differences on the outcome measurements.

DETAILED DESCRIPTION:
Individuals with serious mental illnesses (SMI), as well as those experiencing suicidality or psychiatric crisis encounter police officers frequently in the community. Almost a third of people with SMI have police involved in their pathway to mental health care. Although a variety of strategies to reduce law enforcement involvement in mental health crisis response are emerging, people with SMI and/or those in crisis will continue to encounter police when officers must serve as first responders, and importantly, during officers' routine patrol duties. As such, officers need training to safely and effectively interact in these situations. The Crisis Intervention Team (CIT) model is a collaborative approach that includes a 40-hour training of officers. CIT has been implemented in thousands of U.S. communities, and some agencies are now mandating all of their officers complete CIT training. Despite widespread support and growing research, a randomized, controlled trial (RCT) has never been conducted to assess the effectiveness of CIT training on officers' actual skills and behaviors. Prior research has relied on officers' self-report of their de-escalation skills and has not directly measured actual performance in a rigorous, standardized, controlled fashion. Furthermore, multi-site studies are lacking, and potential officer-level factors that may moderate CIT training outcomes have yet to be systematically assessed.

This study will partner with six sites across the country representing diverse geographic areas and constituency demographics. There are four Specific Aims of the study. First, the investigators will conduct a rigorous, multisite randomized controlled trial (RCT) of CIT mental health training. Each agency will provide 40 officers, for a total of 240. Among the 40 officers from each agency, half will be randomized to CIT training. Data will be collected using Standardized Scenarios, which will be rated centrally in a blinded fashion (blinded by site, study arm, and time). The primary outcome is actual verbal crisis de-escalation skills / non-verbal physical behavior. Second, the investigators will determine the impact of CIT training on two secondary outcomes: use of procedural justice and disposition-related decision-making.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* English-speaking
* Has not yet taken part in CIT training
* Willing and able to be tested, randomized to CIT training or no training, and re-tested at 3-months and 6-months
* Employment as a police officer from participating site

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Verbal Crisis De-escalation Skills / Non-Verbal Physical Behavior Rating (3 months) | 3 months
  Verbal Crisis De-escalation Skills / Non-Verbal Physical Behavior will be assessed via blinded video ratings. The primary outcome is the total score. Domains include: (1) use of reflective statements, (2) use of summarizing/paraphrasing, (3) labelling of emotions, (4) use of encouraging statements, (5) maintaining a conversational tone, (6) seeking clarification from the subject, (7) speaking in a calm and level voice, (8) displaying empathy, (9) displaying honesty, (10) use of simple instructions, (11) asking directly about suicidal ideation, (12) use of space: maintaining appropriate physical distance from the subject, (13) using cover and objects for safety as appropriate, (14) aspects of body language that promote collaboration. Total score ranges from 0 to 100, with a higher score indicating a better outcome.
Verbal Crisis De-escalation Skills / Non-Verbal Physical Behavior Rating (6 months) | 6 months
  Verbal Crisis De-escalation Skills / Non-Verbal Physical Behavior will be assessed via blinded video ratings. The primary outcome is the total score. Domains include: (1) use of reflective statements, (2) use of summarizing/paraphrasing, (3) labelling of emotions, (4) use of encouraging statements, (5) maintaining a conversational tone, (6) seeking clarification from the subject, (7) speaking in a calm and level voice, (8) displaying empathy, (9) displaying honesty, (10) use of simple instructions, (11) asking directly about suicidal ideation, (12) use of space: maintaining appropriate physical distance from the subject, (13) using cover and objects for safety as appropriate, (14) aspects of body language that promote collaboration. Total score ranges from 0 to 100, with a higher score indicating a better outcome.

SECONDARY OUTCOMES:
Procedural justice | 3 months
  Blinded raters will score procedural justice of participants using a standardized rating scale. The total score will range from 0-100, with a higher score indicating greater procedural justice (better outcome).
Procedural justice | 6 months
  Blinded raters will score procedural justice of participants using a standardized rating scale. The total score will range from 0-100, with a higher score indicating greater procedural justice (better outcome).
Disposition-related decision-making | 3 months
  Participants will report on disposition-related decision-making. The total score will range from 0-100, with a higher score indicating better disposition-related decision-making (better outcome).
Disposition-related decision-making | 6 months
  Participants will report on disposition-related decision-making. The total score will range from 0-100, with a higher score indicating better disposition-related decision-making (better outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Michael T. Compton, MD, MPH, Principal Investigator — Columbia University
Locations (1):
- Columbia University in the CIty of New York, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No